CLINICAL TRIAL: NCT04694131
Title: Task-dependent Effects of TMS on the Neural Biomarkers of Episodic Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10000196; 000196-N
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2023-10-12

CONDITIONS: Normal Physiology
Keywords: Memory performance; Neural Biomarkers; EEG; Noninvasive transcranial magnetic stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer Participants (Other): All participants will receive all conditions and the order of all conditions will be counterbalanced across participants. Statistical comparisons will be within-subjects. There will be two experiment days, during which TMS will be delivered during the behavioral tasks (spatial task trials and encoding phase of the memory task). Participants will receive TMS delivered to parietal cortex on one day and vertex stimulation on the other day. Each experiment day will include one block of TMS delivered prior to task trial onsets and one block delivered simultaneously with trial onsets.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The intervention of interest will be TMS delivered to the region of the left posterior parietal cortex with the greatest connectivity with the left hippocampus derived from the baseline resting-state fMRI session. This region was chosen because of its dense connections with the hippocampus, allowing stimulation of this location to modulate function of the hippocampal-cortical network. The control intervention target will be vertex, a commonly used active control site which does not influence neural or behavioral activity.

SUMMARY:
Background:

Transcranial magnetic stimulation (TMS) of the brain has been used to change the activity and connections in the brain to improve memory. Researchers are interested in how these brain changes cause memory improvements and how activity at the time of stimulation may change the effects of TMS.

Objective:

To learn how brain stimulation can be used to improve memory.

Eligibility:

Healthy adults ages 18-40

Design:

Participants will be screened with a medical record review.

Participants will have 3 study visits.

At visit 1, participants will have a physical exam and will talk about their health. They will have magnetic resonance imaging (MRI). The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, participants will lie on a table that can slide in and out of the scanner. A coil will be placed over the head. Participants will be asked to keep their eyes focused on a small cross on a computer screen inside the scanner. The scanner makes loud noises. Participants will get earplugs.

At visits 2 and 3, participants will have TMS and perform tasks. For TMS, a wire coil encased in plastic is held on the scalp. When the coil is triggered, a brief electrical current passes through the coil and creates a magnetic pulse that stimulates the brain. During TMS, an electroencephalogram (EEG) will record brain activity. For the EEG, a cloth cap with electrodes is fitted on the participant s head. Participants will complete a memory task and a spatial processing task. They will also complete surveys about their mental state.

Participation will last 2-3 weeks.

DETAILED DESCRIPTION:
Study Description:

The Behavioral Neurology Unit studies the human brain systems underlying learning and adaptation with the goal of finding interventions to make these processes more efficient. In this study, we are interested in examining how the task state of the episodic memory network influences the effect of faciliatory TMS on memory and its EEG neural correlates. It is hypothesized that Network-targeted parietal-TMS will improve memory performance and enhance EEG biomarkers of successful memory performance, but that these changes will be modulated by the ongoing task activity during stimulation.

Objectives:

Primary Objectives:

Investigate how TMS modulates EEG neural measures of successful memory and the association of this modulation with behavioral performance

Examine how memory task state influences susceptibility to plasticity via TMS and determine the optimal neural state for improving memory

Exploratory Objectives:

Search for MRI predictors of the effects of TMS

Endpoints:

Primary Endpoints: Memory performance, Late Positive Posterior ERP, evoked theta/alpha power (secondary), EEG functional connectivity (secondary)

Exploratory Endpoints: fMRI resting state functional connectivity, fractional anisotropy

ELIGIBILITY:
INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Ability of subject to understand and the willingness to sign a written informed consent document.
3. Age 18-40 (inclusive)

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any current major neurological or psychiatric disorder such as (but not limited to) stroke, Parkinson disease, Alzheimer disease, schizophrenia or major depression
2. History of seizure
3. Medications acting on the central nervous system, such as those that lowers the seizure threshold such as neuroleptics, beta lactams, isoniazid, metronidazole; benzodiazepines, tricyclic or other antidepressants; or prescription stimulants.
4. Inability to provide informed consent
5. Ferromagnetic metal in the cranial cavity or eye, implanted neural stimulator, cochlear implant, or ocular foreign body
6. Implanted cardiac pacemaker or auto-defibrillator or pump
7. Non-removable body piercing
8. Claustrophobia
9. Inability to lie supine for 1 hour
10. Pregnancy, or plans to become pregnant during the study.
11. Members of the NINDS BNU
12. Subjects who have contraindications to MRI will follow the NMR Center guidelines for MR safety.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It has not been determined if it is beneficial or feasible to share IPD. This will be decided at a later time.

REFERENCES:
- [Background] Hermiller MS, Chen YF, Parrish TB, Voss JL. Evidence for Immediate Enhancement of Hippocampal Memory Encoding by Network-Targeted Theta-Burst Stimulation during Concurrent fMRI. J Neurosci. 2020 Sep 9;40(37):7155-7168. doi: 10.1523/JNEUROSCI.0486-20.2020. Epub 2020 Aug 17. PMID 32817326
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Silvanto J, Bona S, Cattaneo Z. Initial activation state, stimulation intensity and timing of stimulation interact in producing behavioral effects of TMS. Neuroscience. 2017 Nov 5;363:134-141. doi: 10.1016/j.neuroscience.2017.09.002. Epub 2017 Sep 8. PMID 28893648
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000196-N.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the NIH healthy volunteer database and the NIH postbac list serve, as well as individuals who self-referred. Recruitment of study participants occurred from July 2021 to February 2023.
Pre-assignment Details: 43 participants were consented to the study and 32 participants successfully completed all study requirements.
Groups:
- Healthy Participants: Healthy participants undergoing all study procedures
Period: Overall Study
Arm/Group | Healthy Participants
Started | 43
Completed | 32
Not Completed | 11
Not completed — Withdrawal by Subject | 7
Not completed — Screen Failure | 1
Not completed — High stimulation threshold | 3

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Memory Performance
Description: Participants completed a memory task with simultaneous EEG acquisition and transcranial magnetic stimulation (TMS) delivered to either a memory-relevant parietal lobe target or a vertex control site. Participants were shown a series of objects in one of four quadrants on the screen, with TMS delivered either prior to or concurrent with the trial onset. They were instructed to remember the object and the location. This outcome measure examines the accuracy of memory for the item and the location (context), presented as the percentage of successful trials. Accuracy is shown for each stimulation condition (parietal or vertex location, before or during the trial)
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: proportion accuracy
Groups:
- Item: Memory for item recognition
- Context: Memory for spatial location of item
Arm/Group | Item | Context
Number analyzed (Participants) | 32 | 32
proportion accuracy
  Parietal, before TMS | 0.89 (0.01) | 0.64 (0.03)
  Parietal, during TMS | 0.91 (0.01) | 0.66 (0.03)
  Vertex, before TMS | 0.92 (0.01) | 0.69 (0.02)
  Vertex, during TMS | 0.89 (0.01) | 0.66 (0.03)

2. Primary Outcome: Late Positive Posterior (ERP) Event Related Potential
Description: Participants completed a memory task with simultaneous EEG acquisition and transcranial magnetic stimulation (TMS) delivered to either a memory-relevant parietal lobe target or a vertex control site. Participants were shown a series of objects in one of four quadrants on the screen, with TMS delivered either prior to or concurrent with the trial onset. They were instructed to remember the object and the location. This outcome measure examines the neural response to trials which were later remembered relative to trials which were later forgotten. Values represent the difference in average EEG amplitude, in uV, between remembered and forgotten trials and compared across each stimulation condition (parietal or vertex location, before or during the trial)
Time Frame: During encoding (with TMS) and during retrieval (after TMS)
Population: Due to EEG trigger issues, only 14 subjects were able to complete the retrieval arm and have data analyzed as ERPs.
Measure: Mean (Standard Deviation); unit: uV
Groups:
- Encoding: ERP amplitude during encoding (uV)
- Retrieval: ERP amplitude during retrieval (uV)
Arm/Group | Encoding | Retrieval
Number analyzed (Participants) | 32 | 14
uV
  Parietal, before TMS | 1.49 (0.83) | -0.11 (1.47)
  Parietal, during TMS | 1.43 (0.63) | 1.29 (1.88)
  Vertex, before TMS | 0.96 (0.76) | -0.91 (1.35)
  Vertex, during TMS | -1.07 (1.41) | 0.79 (2.16)

3. Secondary Outcome: Theta/Alpha Power
Description: Participants completed a memory task with simultaneous EEG acquisition and transcranial magnetic stimulation (TMS) delivered to either a memory-relevant parietal lobe target or a vertex control site. Participants were shown a series of objects in one of four quadrants on the screen, with TMS delivered either prior to or concurrent with the trial onset. They were instructed to remember the object and the location. This outcome measure examines the neural response to trials which were later remembered relative to trials which were later forgotten. Values represent the difference in average task-evoked power in the theta/alpha range (4-13Hz), in uV, between remembered and forgotten trials and compared across each stimulation condition (parietal or vertex location, before or during the trial)
Time Frame: During encoding (with TMS) and during retrieval (after TMS)
Population: Due to EEG trigger issues, only 14 subjects had retrieval data analyzed as task-evoked power
Measure: Mean (Standard Deviation); unit: uV
Groups:
- Encoding: Theta/alpha power during encoding (uV)
- Retrieval: Theta/alpha power during retrieval (uV)
Arm/Group | Encoding | Retrieval
Number analyzed (Participants) | 32 | 14
uV
  Parietal, before trial TMS | 1.46 (2.29) | -0.18 (0.56)
  Parietal during trial TMS | 0.94 (3.20) | 0.06 (0.46)
  Vertex, before trial TMS | 2.25 (5.04) | 0.18 (0.50)
  Vertex, during trial TMS | 1.07 (3.50) | -0.06 (0.56)

ADVERSE EVENTS:
Time Frame: During and Immediately after TMS session
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04694131/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04694131/ICF_001.pdf